CLINICAL TRIAL: NCT07341971
Title: Effect of Non-invasive Vagal Nerve Stimulation on Selected Outcomes in Central Obesity
Acronym: NVN-CO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Lamiaa Zakaria Abd El Salam Salama, Assistant lecturer, Faculty of physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/006137
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- auricular vagus stimulation (Experimental): Transcutanous Electrial Nerve Stimulation
  Interventions: Device: Transcutanous Auricular vagus nerve stimulation
- Sham (Sham Comparator): Sham Stimulation
  Interventions: Device: Sham

INTERVENTIONS:
Device: Transcutanous Auricular vagus nerve stimulation — Non-invasive Auricular Vagus Stimulation
  Arms: auricular vagus stimulation
Device: Sham — Non working device
  Arms: Sham

SUMMARY:
Trans Cutanous Electric Nerve Stimulation of Auricular Vagus Nerve

ELIGIBILITY:
Inclusion Criteria:

* Sixty male
* Age ranges from 18 to 35
* All them are medically stable with no chronic disease
* waist circumference more than 90

Exclusion Criteria:

* Individuals with metabolic diseases
* Individuals taking cholesterol lowering drugs, Anti-hypertensive drugs, Oral-hypoglycemic drugs
* smokers

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-05-25 (Estimated); Study Completion 2026-05-25 (Estimated)

PRIMARY OUTCOMES:
Change in serum Interleukin-6 (IL-6) | Baseline and after 8 weeks of intervention
  serum Interleukin-6 levels will be measured using (ELIZA)

SECONDARY OUTCOMES:
Waist Circumference | Baseline and after 8 weeks of intervention
  Measurement of waist circumference in centimeters as an indicator of central adiposity
Body Shape Index (ABSI) | Baseline and after 8 weeks of intervention
  Assessment of body shape using A Body Shape Index calculated from waist circumference, height, and weight.
Depression Anxiety Stress Scale (DASS-21) Score | Baseline and after 8 weeks of intervention
  Evaluation of psychological status including depression, anxiety, and stress using the validated Depression Anxiety Stress Scale
  -21 questionnaire Higher scores indicate greater severity of emotional state The total score represents the sum of all 21 items multiplied by two. Sub scale scores for depression, anxiety and stress will be calculated and analyzed separately.
Pittsburgh Sleep Quality Index (PSQI) | Baseline and after 8 weeks of intervention
  Assessment of sleep quality using the Pittsburgh Sleep Quality Index questionnaire.
  The total score ranges from 0 to 21 Score greater than 5 indicate poor sleep quality.
Gut Feeling Questionnaire Score | Baseline and after 8 weeks of intervention
  Evaluation of gut-related symptoms and gut-brain interaction using a gut feeling questionnaire The total score is calculated by summing all questionnaire items, with higher scores indicating worse gut feelings.

CONTACTS AND LOCATIONS:
Overall Officials: Nessreen G Al-Nahas, Professor, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared